CLINICAL TRIAL: NCT01211834
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study of the Efficacy and the Safety During Treatment With Tocilizumab vs Placebo in Combination With Traditional DMARD Therapy in Patients With Moderate to Severe Active RA and an Inadequate Response to Current DMARD Therapy
Brief Title: Efficacy and Safety of Tocilizumab in Combination With DMARDs in Patients With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Professor. Young-Wook song, Seoul National Univ. Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CWP-TCZ301
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Antirheumatic Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tocilizumab 8mg/kg+DMARDs (Experimental)
  Interventions: Drug: tocilizumab; Drug: DMARDs
- Placebo+DMARDs (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: DMARDs

INTERVENTIONS:
Drug: tocilizumab — intravenously at dose of 8mg/kg over 1 hour infusion every 4weeks
  Arms: Tocilizumab 8mg/kg+DMARDs
Drug: DMARDs — Methotrexate(MTX) and/or 1 DMARDs(chloroquine, hydroxychloroquine, parenteral gold, sulfasalazine, azathioprine, and leflunomide)
  Arms: Tocilizumab 8mg/kg+DMARDs
Drug: Placebo — intravenously over 1 hour infusion every 4weeks
  Arms: Placebo+DMARDs
Drug: DMARDs — Methotrexate(MTX) and/or 1 DMARDs
  Arms: Placebo+DMARDs

SUMMARY:
The purpose of this study is to assess the efficacy and safety of tocilizumab vs placebo, in combination with stable, ongoing therapy, with regard to reduction in signs and symptoms in patients with moderate to severe active RA and inadequate response to current DMARD treatment

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >= 18 years of age
* Active RA of > 6monts duration
* Received permitted DMARDs each at a stable dose for at least 8 weeks

Exclusion Criteria:

* Rheumatic autoimmune disease other than RA
* Significant systemic involvement secondary to RA
* ALT or AST > ULNⅹ1.5
* Platelet count < 100,000/mm3
* Hemoglobin < 8.5 g/dL
* White blood cells < 3,000/mm3
* Absolute neutrophil count < 2,000/mm3
* Absolute lymphocyte count < 500/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with ACR20 responses | 24weeks
  Proportion of patients with ACR20 responses at post therapy

SECONDARY OUTCOMES:
Proportion of patients with ACR50 and ACR70 responses at post therapy | 24weeks
Change of DAS28, HAQ, individual parameter in ACR core set, hemoglobin | 24weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National Univ. Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Choi IA, Sagawa A, Lee EY, Lee EB, Song YW. Tocilizumab Increases Body Weight and Serum Adipokine Levels in Patients with Rheumatoid Arthritis Independently of Their Treatment Response: a Retrospective Cohort Study. J Korean Med Sci. 2020 Jun 8;35(22):e155. doi: 10.3346/jkms.2020.35.e155. PMID 32508063